CLINICAL TRIAL: NCT02417246
Title: Open-Labeled Pharmacokinetic and Pharmacodynamic (PK-PD) Studies of Metoprolol ER
Brief Title: Open-Labeled PK-PD Studies of Metoprolol ER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201500092; FD14-024 (Other Grant/Funding Number: US FOOD AND DRUG ADMN); OCR15985 (Other: Universiy of Florida)
Record Dates: First submitted 2015-04-01; First posted 2015-04-15 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Blood Pressure
Keywords: pharmacokinetics; pharmacodynamics; pharmacogenetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Sequence A (Active Comparator): Start with brand name metoprolol ER, switch to Generic B metoprolol, switch back to brand name metoprolol ER, then switch to Generic A metoprolol
  Interventions: Drug: brand name metoprolol ER; Drug: Generic A; Drug: Generic B
- Study Sequence B (Active Comparator): Start with brand name metoprolol ER, switch to Generic A metoprolol, switch back to brand name metoprolol ER, then switch to Generic B metoprolol.
  Interventions: Drug: brand name metoprolol ER; Drug: Generic A; Drug: Generic B

INTERVENTIONS:
Drug: brand name metoprolol ER — This medication will be taken for 7 to 28 days
  Other Names: Metoprolol extended-release (ER)
Drug: Generic A — This medication will be taken for 7 days
  Other Names: Metoprolol extended-release (ER)
Drug: Generic B — This medication will be taken for 7 days
  Other Names: Metoprolol extended-release (ER)

SUMMARY:
Recently, the quality of generic metoprolol extended-release (ER) products has been called into question with reports of inconsistent effects when switching from the brand name product to a generic formulation. Problems with how the body processes these drugs could have serious and widespread consequences given the high frequency of metoprolol ER use in the management of various cardiovascular disorders, including high blood pressure, coronary heart disease, heart failure, and cardiac arrhythmias. Investigators hypothesize that both product- and subject-specific factors lead to variability in the way the body breaks down the drug (pharmacokinetics) and clinical response to generic versus name brand metoprolol ER formulations. Investigators will study the brand name and generic metoprolol ER formulations in subjects with high blood pressure to compare the pharmacokinetics and cardiovascular responses among equivalent labeled doses of each product (brand name and two approved generics).

The study objective is to provide information on how the body breaks down generic and brand name metoprolol ER products (pharmacokinetics) and how the body responds to generic and brand name metoprolol ER products (pharmacodynamics) to better understand if generic metoprolol ER products are as good as the brand name product.

DETAILED DESCRIPTION:
As a participant in this study the following will happen.

A study nurse will draw 3 teaspoonfuls (15 ml) of blood. Two teaspoons (10ml) will be drawn for basic blood work and one teaspoon (5ml) will be drawn for genotyping. The study physician will perform a physical exam and discuss all medical history.

The study will be randomized to one of two groups like flipping a coin.

* Study Sequence A- start with brand name metoprolol ER, switch to Generic B metoprolol, switch back to brand name metoprolol ER, then switch to Generic A metoprolol
* Study Sequence B- start with brand name metoprolol ER, switch to Generic A metoprolol, switch back to brand name metoprolol ER, then switch to Generic B metoprolol.

Each study sequence will consist of treatment with brand name metoprolol ER for 2 periods, treatment with Generic A metoprolol ER for one period, and treatment with Generic B metoprolol ER for one period. The generic drug periods will be in a different order for each study group. During the times the switch will take place the following tests will be performed: 24-hour pharmacokinetic parameter assessment, 24-hour heart rate monitoring, 24-hour blood pressure monitoring, 24-hour holter monitoring, exercise treadmill to induce heart rate, and a 24-hour gastric potential hydrogen (pH) monitoring via a wireless capsule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be targeted for enrollment based on current treatment of their hypertension with a beta-blocker or known tolerability to a beta-blocker based on their previous participation in the Pharmacogenomic Evaluation of Antihypertensive Responses studies (PEAR-1 and PEAR-2). If necessary to meet enrollment targets, additional patients will be recruited from the existing patient population in the University of Florida Health Family Medicine clinic or through other means.

Exclusion Criteria:

* Documented secondary forms of hypertension
* Known cardiovascular disease (including history of angina pectoris, myocardial infarction, coronary revascularization procedure, heart failure, or presence of a cardiac pacemaker)
* Known cerebrovascular disease (including stroke and TIA)
* Known peripheral vascular disease
* Diabetes mellitus (Type 1 or 2) (defined as a diabetes diagnosis in the medical record or fasting blood glucose greater than or equal to 126 mg per dl or nonfasting blood glucose greater than or equal to 200 mg per dl on screening laboratories)
* Systolic blood pressure (SBP) greater than180 mm Hg on screening visit
* Heart rate less than 55 bpm on screening visit (in the absence of treatment with a beta-blocker)
* Renal insufficiency (serum creatinine greater than 1.5 in men or greater than 1.4 in women on screening laboratories)
* Liver enzymes (ALT and or AST) greater than 3 times the upper limit of normal on screening laboratories.
* Known Raynaud's phenomenon
* Known asthma or chronic obstructive pulmonary disease
* Pregnancy or lactation
* Gastric bezoar
* Swallowing disorders
* Strictures
* Fistulas
* GI obstruction
* Severe dysphagia
* Crohn's disease
* Diverticulitis
* Any implantable electromedical device
* Use of non-dihydropyridine calcium channel blockers (diltiazem or verapamil)
* Use of digoxin to avoid additive effects on heart rate

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Cavallari, PharmD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Family Medicine at Hampton Oaks Medical Plaza, Gainesville, Florida
  - Oak Hammock at the University of Florida, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 participants were consented with 10 participants as screen fails, 2 declining to further participate, and 1 unable to fit standard monitoring equipment.
Groups:
- Sequence A: Brand name metoprolol ER for 7 to 28 days, and then switch to generic B metoprolol for 7 days, Brand name metoprolol ER for 7 to 28 days, generic A metoprolol for 7 days
- Sequence B: Brand name metoprolol ER for 7 to 28 days, and then switch to generic A metoprolol for 7 days, Brand name metoprolol ER for 7 to 28 days, generic B metoprolol for 7 days
Period: Phase 1 Brand Name Metoprolol ER
Arm/Group | Sequence A | Sequence B
Started | 24 | 24
Completed | 20 | 20
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3
Period: Phase 2 1st Generic Administered
Arm/Group | Sequence A | Sequence B
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Phase 3 Brand Name Metoprolol ER #2
Arm/Group | Sequence A | Sequence B
Started (One patient completed Phase 2 but did not start Phase 3. His data were included in analysis.) | 19 | 20
Completed | 18 | 20
Not Completed | 1 | 0
Period: Phase 4 2nd Generic Administered
Arm/Group | Sequence A | Sequence B
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 18 participants who were administered both brand name metoprolol ER and Generic B and 18 participants who were administered both brand name metoprolol ER and Generic A were analyzed
Groups:
- Sequence A: Brand Name Metoprolol ER and Generic B: This group will start with the brand name metoprolol ER for 7 to 28 days, and then switch to Generic B metoprolol for 7 days.
  Brand name metoprolol ER: This medication will be taken for 7 to 28 days
  Generic B metoprolol: This medication will be taken for 7 days
  Generic A metoprolol: This medication will be taken for 7 days
- Sequence B: Brand Name Metoprolol ER and Generic A: This group will start with the brand name metoprolol ER for 7 to 28 days, and then switch to Generic A metoprolol for 7 days.
  Brand name metoprolol ER: This medication will be taken for 7 to 28 days
  Generic A metoprolol: This medication will be taken for 7 days
  Generic B metoprolol: This medication will be taken for 7 days
- Total: Total of all reporting groups
Arm/Group | Sequence A: Brand Name Metoprolol ER and Generic B | Sequence B: Brand Name Metoprolol ER and Generic A | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 18 subjects who were administered both brand name metoprolol ER and Generic A; and 18 subjects who were administered both brand name metoprolol ER and Generic B were analyzed
  years | 55 (11) | 51 (12) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 18 subjects who were administered both brand name metoprolol ER and Generic B and 18 subjects who were administered both brand name metoprolol ER and Generic A were analyzed
  Participants
    Female | 9 | 8 | 17
    Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30 (4) | 31 (5) | 30 (5)
Weight [Mean (Standard Deviation); unit: kg] | 85 (15) | 93 (23) | 89 (20)
Height [Mean (Standard Deviation); unit: cm] | 169 (10) | 172 (12) | 171 (11)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: The AUC of Brand name metoprolol ER will be compared against each generic for determination of bioequivalence. The mean and standard deviation (SD) values of AUC are entered separately for the 50mg, 100mg and 150mg doses. Results are reported for brand name metoprolol ER, Generic B and Generic A.
Time Frame: 0.0, 0.30, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 20.0, 24.0 hours post dose
Population: This is a 2-way crossover analysis
Measure: Mean (Standard Deviation); unit: ng.hr/ml
Units Other Than Participants: Plasma
Groups:
- Brand Name Metoprolol ER: Brand name metoprolol ER received in Phase 1
- Generic B: Generic B received in Phase 2 or Phase 4
- Generic A: Generic A received in Phase 2 or Phase 4
Arm/Group | Brand Name Metoprolol ER | Generic B | Generic A
Number analyzed (Participants) | 36 | 35 | 35
Number analyzed (Plasma) | 36 | 35 | 35
ng.hr/ml
  50mg | 645.5 (461.4) | 633.0 (523.2) | 654.0 (446.0)
  100mg | 1584.4 (671.1) | 1446.8 (604.3) | 1492.3 (393.3)
  150mg | 12176.1 (7686.6) | 12790.2 (0) | 9926.6 (4383.9)
Statistical Analysis 1: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A paired t-test was used to compare mean values of AUC0-24 for brand name metoprolol ER and Generic B at the 50mg dose. With a sample size of 38, at an alpha level of 0.025 (0.05/2 comparisons), using a 2-sided paired t test, we would have >80% power to detect a 16% difference in AUC; p = 0.3, t-test, 2 sided; Average AUC from 0 to 24 hours (0-24) for patients on the 50mg dose of brand name metoprolol ER and Generic B were compared by a paired t-test (n=28); Mean Difference (Final Values) = 45.1, 95% CI 2-sided [-41.1 to 131.2], Standard Deviation 222.2
Statistical Analysis 2: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A bioequivalence (BE) test was performed for patients who were administered the 50mg dose. BE was declared if 90% confidence interval for the ratio of the population geometric means of the AUC0-24 for Generic B to brand name metoprolol ER falls within 0.8 to 1.25; The analysis included a total of 20 patients on Generic B and brand name metoprolol ER, which is less than the initial plan of including 38 patients; Geometric mean ratio = 0.85, 90% CI 2-sided [0.76 to 0.95]
Statistical Analysis 3: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A paired t-test was used to compare mean values of AUC0-24 for brand name metoprolol ER and Generic A at the 50mg dose. With a sample size of 38, at an alpha level of 0.025 (0.05/2 comparisons), using a 2-sided paired t test, we would have >80% power to detect a 16% difference in AUC; p = 0.8, t-test, 2 sided; Average AUC0-24 for patients on the 50mg dose who were administered brand name metoprolol ER and Generic A were compared using a paired t-test (n=29); Mean Difference (Final Values) = 7.2, 95% CI 2-sided [-60.0 to 74.3], Standard Deviation 176.5
Statistical Analysis 4: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A bioequivalence (BE) test was performed for patients who were administered the 50mg dose. BE was declared if the 90% confidence interval for the ratio of the population geometric means of the AUC0-24 for Generic A to brand name metoprolol ER fell within 0.8 to 1.25; This analysis included 21 individuals who were administered brand name metoprolol ER and Generic A, which is less than the initial plan of including 38 patients; Geometric mean ratio = 0.93, 90% CI 2-sided [0.86 to 1.01]

2. Primary Outcome: Peak Plasma Concentration (Cmax) of Metoprolol Succinate
Description: The Peak Plasma Concentration (Cmax) of Brand name metoprolol ER will be compared against each generic for determination of bioequivalence. The mean and SD values of Cmax are entered separately for the 50mg, 100mg and 150mg doses. Results are reported for brand name metoprolol ER, Generic B and Generic A.
Time Frame: 0.0, 0.30, 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 16.0, 20.0, 24.0 hours post dose
Population: A two-way cross over study in which patients are administered brand name metoprolol ER and Generic B or Generic A
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brand Name Metoprolol ER | Generic B | Generic A
Number analyzed (Participants) | 36 | 35 | 35
ng/mL
  50mg | 36.6 (24.0) | 35.0 (26.9) | 39.9 (22.9)
  100mg | 87.8 (33.3) | 76.5 (31.3) | 83.0 (20.9)
  150mg | 653.3 (399.8) | 613.8 (87.1) | 477.0 (193.7)
Statistical Analysis 1: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A paired t-test was used to compare the mean values of Cmax for brand name metoprolol ER and Generic B at the 50mg dose. With a sample size of 38, at an alpha level of 0.025 (0.05/2 comparisons), using a 2-sided paired t-test, we would have >80% power to detect a 11% difference in Cmax; p = 0.2, t-test, 2 sided; Average Cmax for patients on the 50mg dose who were administered brand name metoprolol ER and Generic B were compared using a paired t-test (n=29); Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-1.5 to 6.6], Standard Deviation 10.7
Statistical Analysis 2: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A bioequivalence (BE) test was performed for patients who were administered the 50mg dose. BE was declared if the 90% confidence interval for the ratio of the population geometric means of Cmax for Generic B to brand name metoprolol ER fell within 0.8 to 1.25; The analysis included a total of 29 patients on Generic B and brand name metoprolol ER, which is less than the initial plan of including 38 patients; Geometric mean ratio = 0.87, 90% CI 2-sided [0.79 to 0.95]
Statistical Analysis 3: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A paired t-test was used to compare the mean values of Cmax for brand name metoprolol ER and Generic A at the 50mg dose. With a sample size of 38, at an alpha level of 0.025 (0.05/2 comparisons), using a 2-sided paired t-test, we would have >80% power to detect a 11% difference in Cmax; p = 0.3, t-test, 2 sided; Average Cmax for patients on the 50mg dose who were administered brand name metoprolol ER and Generic A were compared using a paired t-test (n=29); Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-7.3 to 2.3], Standard Deviation 12.6
Statistical Analysis 4: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A bioequivalence (BE) test was performed for patients who were administered the 50mg dose. BE was declared if the 90% confidence interval for the ratio of the population geometric means of Cmax for Generic A to brand name metoprolol ER fell within 0.8 to 1.25; The analysis included a total of 29 patients on Generic A and brand name metoprolol ER, which is less than a pre-planned sample size of 38; Geometric mean ratio = 1.12, 90% CI 2-sided [1.02 to 1.23]

3. Secondary Outcome: The Heart Rate Variability (HRV) Response to Brand Name Metoprolol ER Versus Each Generic Formulation of Metoprolol Succinate.
Description: 24-h digital heart rate monitor analyses were obtained after Phase 1 (brand name metoprolol ER ), Phase 2 (Generic B or Generic A), and Phase 4 (Generic A or Generic B). Data were analyzed by quartiles. One 5-minute epoch from each hour of each quartile was selected based on absence of a significant number of ectopic beats and artifact from which spectral measures were calculated: high-frequency variability (measure of parasympathetic activity), low-frequency variability (measure of sympathetic activity). The ratio of low-to-high frequency variability was calculated for each quartile. The averages of values obtained for each hour of each quartile constituted the final quartile measures that were used for analysis. The low to high frequency ratio obtained for each quartile represents the balance between sympathetic and parasympathetic nervous system activity and was the primary variable for heart rate variability analysis.
Time Frame: Heart rate variability (Low-to-High Frequency Ratio) over each quartile of 6 hours in the 24-hr period
Population: The analysis aimed to compare HRV (Low-to-High Frequency Ratio) for patients who took Brand name metoprolol ER and a generic formulation (Generic B or Generic A). Low to High Frequency Ratio values are entered for each quartile for Brand name metoprolol ER, Generic B and Generic A
Measure: Mean (Standard Deviation); unit: no units
Arm/Group | Brand Name Metoprolol ER | Generic B | Generic A
Number analyzed (Participants) | 36 | 35 | 35
no units
  Low to High Frequency Ratio: Quartile1 | 2.08 (2.43) | 1.67 (1.21) | 1.79 (1.06)
  Low to High Frequency Ratio: Quartile 2 | 2.06 (1.74) | 1.64 (1.05) | 1.95 (1.50)
  Low to High Frequency Ratio: Quartile 3 | 2.06 (1.57) | 1.92 (1.21) | 2.08 (0.99)
  Low to High Frequency Ratio: Quartile 4 | 1.95 (1.18) | 2.22 (1.79) | 2.34 (1.73)
Statistical Analysis 1: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A mixed effect model for repeated measures was used to model medication effect on HRV comparing brand name metoprolol ER to Generic B, adjusting for quartile, (quartile*med) interaction, and treatment assignment; p = 0.0858, Mixed Models Analysis; Slope = -0.7, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A mixed effect model for repeated measures was used to model medication effect on HRV comparing brand name metoprolol ER to Generic A, adjusting for quartile,(quartile*med) interaction, and treatment assignment; p = 0.0168, Mixed Models Analysis; Slope = -0.6, Standard Error of Mean 0.3 — p for medication*quartile interaction considered significant if p<0.025

4. Secondary Outcome: Blood Pressure Values (Systolic and Diastolic) Compared Between Brand Name Metoprolol ER and Each Generic Metoprolol Formulation (Generic B, Generic A)
Description: 24-hr ambulatory blood pressure (BP) recordings taken 4 times per hour (every 15 minutes) between 6AM and 11PM and 2 times per hour (every 30 minutes) 11PM and 6AM were obtained after Phase 1 (Brand name metoprolol ER), Phase 2 (Generic B or Generic A), and Phase 4 (Generic A or Generic B).
Time Frame: Average value over each quartile of 6 hours in the 24-hr period
Population: The analysis aimed to compare mean BP values in Hg mm between the brand name and each of the generic (Generic B or Generic A) formulation of metoprolol succinate. Patients were included in the analysis if they took brand name metoprolol ER and at least one generic.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Brand Name Metoprolol ER | Generic B | Generic A
Number analyzed (Participants) | 36 | 35 | 35
mm Hg
  Systolic Blood Pressure: quartile 1 | 132.8 (14.1) | 129.6 (15.0) | 129.1 (15.1)
  Systolic Blood Pressure: quartile 2 | 134.1 (16.0) | 131.3 (16.1) | 131.0 (16.4)
  Systolic Blood Pressure: quartile 3 | 124.1 (17.2) | 121.0 (16.3) | 123.1 (15.6)
  Systolic Blood Pressure: quartile 4 | 129.3 (16.6) | 127.7 (17.0) | 128.0 (15.8)
  Diastolic Blood Pressure: quartile 1 | 80.8 (10.5) | 79.3 (10.2) | 78.3 (11.1)
  Diastolic Blood Pressure: quartile 2 | 80.8 (11.6) | 80.3 (11.4) | 78.5 (11.7)
  Diastolic Blood Pressure: quartile 3 | 75.4 (13.2) | 73.2 (11.4) | 74.4 (10.4)
  Diastolic Blood Pressure: quartile 4 | 79.2 (10.4) | 80.0 (13.3) | 78.1 (9.6)
Statistical Analysis 1: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour ambulatory systolic blood pressure (SBP) by quartile for 35 patients receiving brand name metoprolol ER and Generic B; p = 0.203, Mixed Models Analysis; Slope = -2.39
Statistical Analysis 2: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour ambulatory diastolic blood pressure (DBP) by quartile for 35 patients receiving brand name metoprolol ER and Generic B; p = 0.671, Mixed Models Analysis; Slope = -0.543
Statistical Analysis 3: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour ambulatory SBP by quartile for 35 patients receiving brand name metoprolol ER and Generic A; p = 0.200, Mixed Models Analysis; Slope = -2.371
Statistical Analysis 4: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour ambulatory DBP by quartile for 35 patients receiving brand name metoprolol ER and Generic A; p = 0.068, Mixed Models Analysis; Slope = -2.3290

5. Secondary Outcome: Heart Rate (HR) Response Compared Between Brand Name Metoprolol ER and Each Generic (Generic B, Generic A) Formulation of Metoprolol Succinate
Description: 24-h ambulatory heart rate recordings taken 4 times per hour (every 15 minutes) between 6AM and 11PM and 2 times per hour (every 30 minutes) 11PM and 6AM were obtained after Phase 1 (brand name metoprolol ER), Phase 2 (Generic B or Generic A), and Phase 4 (Generic A or Generic B)
Time Frame: Average value over each quartile of 6 hours in the 24-hr period
Population: The analysis aimed to compare 24-hr HR between the brand name and each generic (generic B or generic A) formulation of metoprolol succinate. Mean and SD values for HR entered for each medication by quartile
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Brand Name Metoprolol ER | Generic B | Generic A
Number analyzed (Participants) | 36 | 35 | 35
bpm
  HR (beats per minute) Quartile one | 65.1 (11.5) | 65.4 (11.5) | 66.1 (11.3)
  HR (beats per minute) Quartile two | 65.3 (11.5) | 65.9 (10.5) | 66.9 (11.5)
  HR (beats per minute) Quartile three | 61.3 (9.9) | 62.8 (10.1) | 63.4 (10.6)
  HR (beats per minute) Quartile four | 61.4 (12.9) | 62.5 (11.6) | 62.5 (11.3)
Statistical Analysis 1: Comparison: Brand Name Metoprolol ER vs Generic B; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour HR by quartile for 35 patients receiving brand name metoprolol ER and Generic B; p = 0.333, Mixed Models Analysis; Slope = 1.233
Statistical Analysis 2: Comparison: Brand Name Metoprolol ER vs Generic A; Test type: Equivalence — A mixed effect model for repeated measures was performed to model the 24-hour HR by quartile for 35 patients receiving brand name metoprolol ER and Generic A; p = 0.368, Mixed Models Analysis; Slope = 1.1340

ADVERSE EVENTS:
Time Frame: Up to 12 weeks since the start of phase one (patients starting their first dose of brand name metoprolol ER)
Description: Safety population included all patients who took at least one dose of study drug (i.e. one dose of brand name metoprolol ER in Phase 1)
Groups:
- Brand Name: Brand Name Metoprolol ER
- Generic A: Generic Metoprolol ER type A
- Generic B: Generic Metoprolol ER type B
Arm/Group | Brand Name | Generic A | Generic B
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 33/48 | 21/38 | 16/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brand Name (N=48) | Generic A (N=38) | Generic B (N=40)
ECG signs of myocardia ischemia (Investigations) | 1 | 0 | 0 — ECG changes observed during stress test. Patient received medical attention and was withdrawn from study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brand Name (N=48) | Generic A (N=38) | Generic B (N=40)
Urinary tract infections (Renal and urinary disorders) | 1 | 0 | 0
Dyspepsia (General disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2
Fatigue (General disorders) | 8 | 2 | 0
Hypertension (Vascular disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 6 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Lower extremity itching and burning
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Sluggishness (General disorders) | 1 | 0 | 0
Hyperhidrosis (General disorders) | 1 | 0 | 0
Syncope (Vascular disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Dyspnoea (Cardiac disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 1 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 1 — 1 mm ST segment depression with quick recovery
Influenza like illness (General disorders) | 1 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Puncture site reaction (Injury, poisoning and procedural complications) | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Pre syncope (Nervous system disorders) | 0 | 0 | 1
Skin burning sensation (Nervous system disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
1. The final study sample size was lower than what was originally proposed based on power analysis.
2. The study protocol did not specify the attainment of steady-state prior to the 24-hour pharmacokinetic and pharmacodynamic studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT02417246/Prot_SAP_ICF_000.pdf